CLINICAL TRIAL: NCT01869192
Title: Differential Gene Regulation During Neoadjuvant Therapy Trial of Epirubicin/Cyclophosphamide (EC) vs Docetaxel/Capecitabine (DX) Regimens in Patients With Large ER-positive and ER-negative Breast Cancers: A Randomized Phase II Trial.
Brief Title: Phase II Trial for Large ER-Negative Breast Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-824.cc
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Malignant Neoplasm of Female Breast
Keywords: Malignant; Neoplasm; Cancer; Female; Breast; Stage II; Stage III
MeSH Terms: conditions — Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Capecitabine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: randomized sequence of therapy.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Arm A: Epirubicin 90 mg/m2 day 1 IV and Cyclophosphamide 600 mg/m2 day 1 IV q 3 weeks for 4 cycles, then surgery, then Docetaxel 75 mg/m2 IV day 1 plus Capecitabine 1000 mg/m2/dose po bid x 14 days q 3 weeks for 4 cycles, then radiation therapy as indicated. Post surgical chemotherapy must be initiated within 35 days after completion of definitive surgical treatment
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Radiation: Radiation Therapy
- Arm B (Active Comparator): Arm B: Docetaxel 75 mg/m2 IV day 1 plus Capecitabine 1000 mg/m2/dose po bid x 14 days q 3 weeks for 4 cycles, then surgery, then Epirubicin 90 mg/m2 day 1 IV and Cyclophosphamide 600 mg/m2 day 1 IV q 3 weeks for 4 cycles, then radiation therapy as indicated. Post surgical chemotherapy must be initiated within 35 days after completion of definitive surgical treatment
  Interventions: Drug: Docetaxel; Drug: Capecitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Epirubicin — Epirubicin 90 mg/m2 d1 q3w
  Other Names: Ellence, Pharmorubicin PFS, Pharmorubicin RDF
  Arms: Arm A
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2 d1 q3w
  Other Names: Cytoxan, Neosar, Cytoxan Lyophilized
  Arms: Arm A
Drug: Docetaxel — Docetaxel 75 mg/m2 d1 q3w
  Other Names: Docefrez, Taxotere
  Arms: Arm B
Drug: Capecitabine — Capecitabine 1000 mg/m2/dose bid x 14d q3w
  Other Names: Xeloda
  Arms: Arm B
Radiation: Radiation Therapy — Standard dosing, fields depending on clinical findings

SUMMARY:
A primary objective of this study is to evaluate the in vivo response of tumor to chemotherapy through gene microarray analysis. Neoadjuvant treatment allows the unique opportunity to observe the in vivo effects of cytotoxic therapy on gene expression in tumor tissue. The investigators plan to evaluate several different questions by comparing gene profiles in different phases of treatment in this study. These are outlined below.

Hypotheses

1. Chemotherapy enriches for tumor cell populations that have enhanced resistance and survival mechanisms. These mechanisms will in part be identifiable through changes in gene expression profiles pre vs. post treatment.
2. Use of two distinct chemotherapy selection pressures, for example a DNA-damaging regimen (epirubicin and cyclophosphamide) or a mitotic spindle/metabolic targeted regimen (docetaxel and capecitabine), will allow for the identification of a smaller set of genes associated to resistance and survival mechanisms of broad importance.
3. Genes associated with enrichment for resistance and survival mechanisms will not be present in large amounts pretreatment in tumors destined for complete pathologic response.

DETAILED DESCRIPTION:
The clinical outcomes of breast cancer treatment are remarkably similar regardless of the regimen used, even though the individual drugs may differ substantially in mechanisms of action. We are interested in identifying a set of genes that may be associated with breast cancer cell survival following selection by chemotherapy. We intend to use two different selection pressures (different chemotherapy regimens with different mechanisms of action) in order to focus on those genes that are regulated similarly in response to either regimen.

Neoadjuvant chemotherapy is in common use for locally advanced breast cancers. Although it does not yet appear to impart a survival advantage, it does enhance the likelihood of breast conserving surgery and also provides important prognostic information. Taxotere appears to add significantly to pathologic complete responses when added to doxorubicin and cyclophosphamide alone. The combination of capecitabine and docetaxel was superior to docetaxel alone in metastatic disease. Many investigators are interested in incorporating this regimen for the treatment of earlier stages of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* The diagnosis of breast cancer can be made by fine-needle aspiration (FNA), core, or tru-cut biopsy. Biopsy must demonstrate invasive adenocarcinoma.
* Patients must have a life expectancy of at least 1 year, excluding their diagnosis of cancer.
* Patients must have a mass on clinical or radiological examination of >1 cm and must be confined to either the breast or to the breast and ipsilateral axilla. Multiple masses permitted, provided one of them is >1cm.
* Patients may enter prior to ER or Her2 status being known, however if Her2 is positive, then the patient is withdrawn from the treatment phase of the trial.
* Patients with palpable mass with distant metastasis and/or palpable supraclavicular lymphadenopathy allowed if definitive local treatment is judged to be necessary.
* Patients may have inflammatory breast cancer.
* Prior to time of entry, patients must have had the following:
* history and physical exam
* blood tests
* chest imaging within the last 3 months (chest x-ray, CT scan, PET/CT)
* bilateral mammogram
* Ultrasound of tumor with placement of clip to localize tumor should it respond completely to chemotherapy is recommended
* Bone scan and MRI of the breast as clinically indicated.
* Patients with clinically palpable lymph nodes are recommended to have a FNA biopsy to document the lymph node status. Patients may undergo a sentinel node biopsy procedure prior to preoperative chemotherapy.
* At time of entry
* White blood cell count (WBC) > 3,000
* platelet count > 100,000
* bilirubin, serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate oxaloacetate transaminase (SGPT), alkaline phosphatase, and serum creatinine must all be < 1.2 x upper limit of normal (ULN)
* calculated creatinine clearance [Cockcroft-Gault] > 50 ml/min. normalized to a 1.73 m2 body surface area (BSA). Patients with benign hyperbilirubinemia are also excluded.
* Patients with bone pain are eligible for inclusion if bone scan and/or roentgenological exam fail to disclose metastatic disease, or if metastatic disease is found, definitive local treatment is to be performed.
* Patients with non-breast malignancies are eligible if they have not received prior chemotherapy, or extensive radiation therapy, and are free from disease for at least two years. Patients with squamous or basal carcinoma of the skin that has been effectively treated, carcinoma in situ of the cervix that has been treated by surgery only are eligible. Patients with prior or simultaneous lobular or ductal carcinoma in situ of the ipsilateral or contralateral breast are also eligible. Patients with bilateral breast cancer for which at least one of the breast cancers meet the eligibility requirements are also eligible.
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of chemotherapy (female patients of childbearing potential).

Exclusion Criteria:

* Patients with Her2 positive breast cancer
* Pregnancy or breast feeding at the time of proposed randomization. Women of childbearing potential with either a positive or no pregnancy test at baseline. Woman of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.
* Prior therapy for this breast cancer.
* Prior chemotherapy for a different breast cancer. Patients who have received prior anthracycline therapy for any malignancy are not eligible.
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the patient from being subjected to any of the treatment options or surgery or would prevent prolonged follow-up.
* Active cardiac disease that would preclude the use of epirubicin. This includes:
* Any documented myocardial infarction or unstable angina;
* Any history of documented congestive heart failure;
* Valvular disease with documented cardiac function compromise;
* Patients with cardiomegaly on chest X-ray, or ventricular hypertrophy on EKG, unless they demonstrate adequate left ventricular ejection fraction (LVEF) > 45% by MUltiple Gated Acquisition (MUGA) or echocardiogram.
* Patients with a cardiac arrhythmia are eligible, provided the arrhythmia is not associated with concomitant heart failure or cardiac dysfunction.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy
* Unwillingness to give written informed consent.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-03-05 (Actual); Primary Completion 2009-12-18 (Actual); Study Completion 2010-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Elias, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: EC Prior to Surgery, Then XT: Arm A: Epirubicin 90 mg/m2 day 1 IV and Cyclophosphamide 600 mg/m2 day 1 IV q 3 weeks for 4 cycles, then surgery, then Docetaxel 75 mg/m2 IV day 1 plus Capecitabine 1000 mg/m2/dose po bid x 14 days q 3 weeks for 4 cycles, then radiation therapy as indicated. Post surgical chemotherapy must be initiated within 35 days after completion of definitive surgical treatment
  Epirubicin: Epirubicin 90 mg/m2 d1 q3w
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 d1 q3w
  Radiation Therapy: Standard dosing, fields depending on clinical findings
- Arm B: XT Prior to Surgery, Then EC: Arm B: Docetaxel 75 mg/m2 IV day 1 plus Capecitabine 1000 mg/m2/dose po bid x 14 days q 3 weeks for 4 cycles, then surgery, then Epirubicin 90 mg/m2 day 1 IV and Cyclophosphamide 600 mg/m2 day 1 IV q 3 weeks for 4 cycles, then radiation therapy as indicated. Post surgical chemotherapy must be initiated within 35 days after completion of definitive surgical treatment
  Docetaxel: Docetaxel 75 mg/m2 d1 q3w
  Capecitabine: Capecitabine 1000 mg/m2/dose bid x 14d q3w
  Radiation Therapy: Standard dosing, fields depending on clinical findings
Period: Preoperative Chemotherapy to Surgery
Arm/Group | Arm A: EC Prior to Surgery, Then XT | Arm B: XT Prior to Surgery, Then EC
Started | 37 | 35
Completed (2 did not go to surgery) | 35 | 34 (one never got treatment on study)
Not Completed | 2 | 1
Not completed — patient choice | 2 | 1
Period: Postoperative Chemotherapy
Arm/Group | Arm A: EC Prior to Surgery, Then XT | Arm B: XT Prior to Surgery, Then EC
Started | 32 (3 did not start postop chemotherapy) | 33
Completed | 32 | 31
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Full Range); unit: years] | 50 [30 to 69] | 50 [33 to 73] | 50 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To describe the overall response rate as measured by physical exam and MRI if indicated using the following definition: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 37 | 35
Participants | 25 | 21

2. Secondary Outcome: Pathological Response
Description: Pathological response (pCR or microscopic only primary) in both primary and nodes using the Miller-Payne criteria for pathologic response.
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 37 | 35
Participants | 2 | 8

ADVERSE EVENTS:
Description: SAE reporting required; AE reporting not required by protocol
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes